CLINICAL TRIAL: NCT05835583
Title: The Effectiveness of the Theory-based Integrated Program on Medication Adherence Among Community-dwelling Patients With Schizophrenia
Brief Title: Theory Based Integrated Program on Medication Adherence Among Community Dwelling Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Principal Investigator, Wen I Liu, Distinguished Professor and Dean, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: The Integrated program
Record Dates: First submitted 2023-01-11; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Schizophrenia; Medication Adherence; Medication Compliance
Keywords: Schizophrenia, Medication Adherence, Randomized control trail,community, schizophrenia
MeSH Terms: conditions — Schizophrenia; Medication Adherence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): Members of the experimental group received routine home visits( by psychiatric mental nurses, and the nurse provided patients with answers to questions about medications or care and handling of life events), and plus a 1-hour theory based integrated program intervention for 12 times in the 1st, 3rd, 5th, 7th, 9th, 11th, 13th, 15th, 17th, 19th, 21st, and 23rd weeks, and each patient received a total of 12 hours of intervention.
  Interventions: Behavioral: The theory based integrated program
- control (No Intervention): The control group received routine home visits by psychiatric mental nurses, and the nurse provided patients with answers to questions about medications or care and handling of life events. The visits and intervention time frequency were the same as those in the experimental group.

INTERVENTIONS:
Behavioral: The theory based integrated program — The theory-based integrated program is administered by a nurse trained in motivational interviewing.In the 12-hour intervention, this program uses motivational interviewing skills to increase the patient's attitude towards medication, enhance the support of significant others around them, and increase the patient's control over their own behavior.
  Arms: experimental

SUMMARY:
This clinical trial aims to evaluate the effectiveness of the theory-based integrated program in promoting medication adherence in patients with schizophrenia. The purpose of this study are:

* To explore the effectiveness of the theory-based integrated program in promoting community-based schizophrenia patients' adherence to medication(like :motivation, attitude and behavior)
* To explore the effectiveness of the theory-based integrated program in improving the psychiatric symptoms of patients with schizophrenia in the community.

Participants (the experimental group) received routine home visits from psychiatric mental nurses, including drug administration, drug side effects and symptom management, life care, and the theory-based program provided by the researcher(treatment as usual + the theory-based integrated program).

The comparison group: received routine home visits from psychiatric mental nurses, including drug administration, drug side effects, and symptom management, life care,(treatment as usual).

DETAILED DESCRIPTION:
Members of the experimental group received routine home visits, plus a 1-hour the theory-based program intervention 12 times in the 1st, 3rd, 5th, 7th, 9th, 11th, 13th, 15th, 17th, 19th, 21st, and 23rd weeks, and each patient received a total of 12 hours of intervention.

The control group received routine home visits by psychiatric mental nurses, and the nurse provided patients with answers to questions about medications or care and handling of life events. The visits and intervention time frequency were the same as those in the experimental group.

Both groups were received baseline (T0), after the 6th hours intervention (T1) and 12th hours intervention by nurses to collect data on the main outcome variables: adherence to medication, mental symptoms, motivation to take medication, and attitude towards medication.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of schizophrenia group, including schizophrenia, affective schizophrenia (schizoaffective disorder);
2. Age between 20 and 64 years old;
3. At least one oral antipsychotic drugs;
4. Living in the community, not participating in day wards, community rehabilitation centers and other rehabilitation institutions on weekdays, no psychiatric outpatient clinics, only home visits by home nurses;
5. Those who can communicate in Chinese and Taiwanese

Exclusion Criteria:

1. Those who have a diagnosis related to organic problems, substance abuse, dementia or mental retardation, and are unable to communicate;
2. Those who have received long-acting injections from the psychiatric department. -

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Medication Adherence Rating Scale；MARS | The time point of measurement is the baseline, the change in the 6th hour after the intervention, and the change in the 12th hour.
  The Medication Adherence Rating Scale(MARS) is a 10-item self-reporting multidimensional instrument describing three dimensions: medication adherence behavior (items 1-4), attitude toward taking medication (items 5-8) and negative side effects and attitudes to psychotropic medication (items 9-10). sponse consistent with non-adherence is coded as 0, whereas a response consistent with adherence is coded as 1. For questions 1-6 and 9-10, a no response is indicative of adherence and is coded as 1, while for questions 7 and 8, a yes response is indicative of adherence and is coded as 1. Total scores on the MARS may range between 0 and 10, with a higher score indicating better medication adherence.
Brief Psychiatric Rating scale；BPRS | The time point of measurement is the baseline, the change in the 6th hour after the intervention, and the change in the 12th hour.
  The Brief Psychiatric Rating scale(BPRS) assesses the level of 18 symptom constructs such as hostility, suspiciousness, hallucination, and grandiosity. It is particularly useful in gauging the efficacy of treatment in patients who have moderate to severe psychoses.Total scores on the MARS may range between 0 and 10, with a higher score indicating better medication adherence.This scale is scored from 0-6, with a total of 16 items, and the total score ranges from 0 to 96. The higher the score, the more obvious the psychiatric symptoms
University of Rhode Island Changed Assessment；URICA | The time point of measurement is the baseline, the change in the 6th hour after the intervention, and the change in the 12th hour.
  The University of Rhode Island Change Assessment Scale (URICA) is a 32 item self-report measure that includes 4 subscales measuring the stages of change: Precontemplation, Contemplation, Action, and Maintenance (there is also a 24 item version). Responses are given on a 5 point Likert scale ranging from (1=strong disagreement to 5=strong agreement),Calculate the score with its calculation formula, and get a score ranging from -2 to 14. The higher the score, the stronger the motivation to change.
Drug Attitude Inventory，DAI-10 | The time point of measurement is the baseline, the change in the 6th hour after the intervention, and the change in the 12th hour.
  The Drug Attitude Inventory(DAI-10) contains six items that a patient who is fully adherent to prescribed medication would answer as 'True', and four they would rate as 'False'. Scores are allocated to each answer and the total score is calculated in the same way as for the DAI-30. The range is -4 to 6 points. The higher the score, the more positive the attitude of taking the medicine, with 0 points as the cut-off point, above 0 means the attitude of taking the medicine is positive; below 0 means the attitude of taking the medicine is negative
Global Assessment of of Functioning, GAF | The time point of measurement is the baseline, the change in the 6th hour after the intervention, and the change in the 12th hour.
  The Global Assessment of Functioning, or GAF, scale is used to rate how serious a mental illness may be. It measures how much a person's symptoms affect their day-to-day life on a scale of 0 to 100.The higher the score, the better the function. A score above 81 means good function, a score below 50 means serious difficulty in function, and a score of 0 means insufficient information

CONTACTS AND LOCATIONS:
Overall Officials: Liu Wen-I, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan